CLINICAL TRIAL: NCT01952106
Title: Effects of Distraction on Pain and Distress During Venepuncture in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201305092RIND
Record Dates: First submitted 2013-09-17; First posted 2013-09-27 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Hospitalism in Children; Pain
Keywords: venepuncture; distraction; distress
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- distraction (Experimental): use the computer game to distract children's pain and anxiety during venepuncture
  Interventions: Other: play computer game

INTERVENTIONS:
Other: play computer game

SUMMARY:
The main purpose of this study is Investigating the effectiveness of distraction by evaluating the children's perception of pain during venepuncture.

ELIGIBILITY:
Inclusion Criteria:

* 5-7 years old
* understanding numeral

Exclusion Criteria:

* mental retard and can not nuderstand numeral

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Visual Analogue pain Scale will be used to evaluate children's pain perception | approximately 15 mins during venepuncture process
  monitor the children's oxygen saturation and pain scale.

CONTACTS AND LOCATIONS:
Overall Officials: chiying Tseng, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan